CLINICAL TRIAL: NCT06927206
Title: Combined Effects of Segmental Vibrator With Neuromuscular Electrical Stimulation for Dorsiflexors on Lower Limb Function in Subacute Stroke
Brief Title: Segmental Vibrator With NMES on Lower Limb Function in Subacute Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC//24/0219 Arooj Shahzad
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Subacute Stroke; Ischemic Stroke
Keywords: Dorsiflexion; FMA; NEMS; Segmental muscle vibrator; Stroke; Spasticity; Vibration
MeSH Terms: conditions — Ischemic Stroke; Stroke; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: assignment
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): Group A: Standard physical therapy and segmental vibrator on dorsiflexor muscle groups
  Interventions: Other: Experimental Group A: Segmental vibrator only on dorsiflexor
- group B (Experimental): Group B: Standard physical therapy and segmental vibrator + electrical stimulation on dorsiflexor muscle group
  Interventions: Other: Experimental Group B: Segmental vibrator + Electrical stimulation on dorsiflexors

INTERVENTIONS:
Other: Experimental Group A: Segmental vibrator only on dorsiflexor — Segmental vibrator only on dorsiflexor:
  After standard physiotherapy session this group received the intervention of segmental vibration. Tibialis anterior muscle targeted for dorsiflexor. The segmental vibration of high frequency i.e 100 Hz and low amplitude (0.2-0.5mm) was applied at muscle belly for 10 min while interpersed with a 1 min break by mean of segmental vibrator.
  Arms: group A
Other: Experimental Group B: Segmental vibrator + Electrical stimulation on dorsiflexors — Segmental vibrator + Electrical stimulation on dorsiflexors:
  After standard physiotherapy session this group received the intervention of neuromuscular electrical stimulations by means of EMS. Two electrodes were used for this procedure. Tibialis anterior muscle targeted for dorsiflexor. One pad of electrode was placed on anterior of lower leg just below tibial tuberisty and other was 5cm below to it .With a 250-microsecond pulse duration, the EMS device was set up to provide a biphasic current with a symmetrical waveform at 50 Hz for 15 seconds. It was also tuned for a 3-second ramp up time and a 30-second rest period. Each respondent set the intensity to the highest level they could tolerate. Secondly, segmental vibrator was applied for focal vibrations on tibialis anterior. The segmental vibration of high frequency i.e 100 Hz and low amplitude (0.2-0.5mm) was applied at muscle belly for 10 min while interpersed with a 1 min break by mean of segmental vibrator.
  Arms: group B

SUMMARY:
Stroke is one of the world's leading causes of death and disability. It can cause a variety of motor disorders, such as apraxia, sensory deficits, abnormal muscle tone, inadequate weight transfer, lack of fine motor skills, incoordination, and balance deficit. These disorders can have a significant negative impact on a person's quality of life.

DETAILED DESCRIPTION:
The definition of a stroke, as given by the World Health Organization (WHO), is a clinical illness that includes focused disruptions in cerebral functioning that develop quickly and have a vascular origin. Cerebrovascular accidents, or strokes, rank third in the world in terms of disability and are the second major cause of mortality. A stroke is a major cause of dementia and depression. A stroke is the abrupt death of some brain cells from a lack of oxygen when blood supply to the brain is interrupted by an artery rupturing or blocking the brain. Across the world, low- and middle-income nations account for 70% of stroke cases and 87% of stroke-related fatalities as well as disability-adjusted life years. Patients who have had a stroke often experience a variety of motor disorders, such as dysphagia and dysarthria, imbalance issues, apraxia, sensory deficiencies, abnormal muscle tone, abnormal motor pattern, inadequate weight transfer, lack of fine motor skills, and muscle weakness. After completing their rehabilitation, 50% to 60% of stroke patients still have some degree of motor impairments, and at least 50% of these patients depend on their daily activities. Muscle paresis and spasticity are two of the most prevalent stroke disabilities.

This study aims to explore the effects of combining focal vibration (FV) with electrical neuromuscular stimulation (NMES) on the ankle dorsiflexors in subacute stroke patients. These techniques are relatively new in neurorehabilitation and have shown promise in reducing muscle stiffness and enhancing movement compared to traditional physiotherapy methods. By focusing on the lower limb issues commonly seen after a stroke, we seek to understand how this combination therapy can improve motor function in these patients. The findings of this study could help in developing more effective treatment strategies for stroke survivors dealing with lower limb dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female patients were included in the study.
* The age range of participants was between 45 and 60 years.
* Participants that were diagnosed with ischemic stroke patient.
* Participants had experienced sub-acute ischemic stroke, specifically 15 days to 12 weeks post-stroke.
* Montreal Cognitive Assessment scores falling within the range of 18-24 were necessary.
* Modified Ashworth scale scores had to be less than +1
* National Institutes of Health Stroke Scale (NIHSS) score falling within the range of 1 to 15 were necessary.
* Participants feel no pain from the vibrator.
* It was anticipated that participants would either be able to give informed consent or have a legal representative who could do so.

Exclusion Criteria:

* People who had a history of serious neurological or mental conditions that would have impeded lower limb motor recovery-aside from stroke-were not included.
* Individuals with severe arthritis or joint injuries, among other illnesses that would have interfered with treatment or evaluations, were not allowed to participate.
* Individuals who had significant hearing or vision impairments that would have hampered treatment or evaluations were not included.
* Individuals undergoing anti-spatial therapy or other clinical trials, those with bilateral brain lesions, and those with ischemic involvement of the cerebellum or basal ganglia were not allowed to participate.
* Participants having metal implants e. g cardiac pacemaker and skin lesion at the site of stimulation electrodes were excluded.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale (for spasticity) | 8 weeks
  The Modified Ashworth Scale (MAS) is a revised version of the original Ashworth Scale that measures spasticity in patients with lesions to the central nervous system. MAS is an assessment that is used to measure the increase in muscle tone. MAS assigns a grade of spasticity from a 0-4 ordinal scale.
Fugl-Meyer Assessment (for lower limb function) | 8 weeks
  Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. The scale is comprised of five domains and there are 155 items in total:
  * Motor functioning (in the upper and lower extremities)
  * Sensory functioning (evaluates light touch on two surfaces of the arm and leg, and position sense for 8 joints)
  * Balance (contains 7 tests, 3 seated and 4 standing)
  * Joint range of motion (8 joints)
  * Joint pain Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform; 1=performs partially; and 2=performs fully. The total possible scale score is 226.
10 Metre Walk Test (mobility) | 8 weeks
  The 10-Metre Walk Test is a performance measure used to assess walking speed in meters per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function. Gait speed is calculated by dividing the total distance to time
Wisconsin Gait Scale (for gait) | 8 weeks
  Wisconsin Gait Scale (WGS) is an observational tool for the evaluation of gait quality in individuals after stroke with hemiplegia. It is divided into four subscales, which assess a total of fourteen spatiotemporal and kinematic parameters of gait observed during the consecutive gait phases.
Goniometer for ROM | 8 weeks
  A goniometer is a valid clinical tool used to measure the range of motion in joints. It used to measure the ankle dorsiflexion ROM.

CONTACTS AND LOCATIONS:
Overall Officials: Aruba Saeed, PhD, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No